CLINICAL TRIAL: NCT02952131
Title: Use of Autologous Adult Adipose-Derived Stem/Stromal Cells in Inflammatory Bowel Disease
Brief Title: Use of Autologous, Adult Adipose-Derived Stem/Stromal Cells in Inflammatory Bowel Disease
Acronym: ADcSVF-IBD
Status: Suspended | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: COVID prevented continuation
Sponsor: Healeon Medical Inc (Industry)
Collaborators: Terry, Glenn C., M.D. (Individual)
Responsible Party: Principal Investigator, Robert W. Alexander, MD, FICS, Principal Investigator, Healeon Medical Inc
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RGV-GARM3
Record Dates: First submitted 2016-10-30; First posted 2016-11-02 (Estimated); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Inflammatory Bowel Diseases
Keywords: IBD,Crohn's,Ulcerative Bowel; Diverticulitis;IBS;UC
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Lipoaspiration Arm 1 (Experimental): Acquisition of Adipose-Derived tissue Stromal Vascular Fraction (AD-tSVF) via closed syringe harvest subdermal fat
  Interventions: Procedure: Lipoaspiration
- AD-cSVF Arm 2 (Experimental): Isolation of cellular stem/stromal cells from subdermal adipose-derived cellular stromal vascular fraction (AD-cSVF)
  Interventions: Procedure: AD-cSVF
- Normal Saline IV Arm 3 (Experimental): Normal Saline IV with AD-cSVF cells
  Interventions: Procedure: Normal Saline IV

INTERVENTIONS:
Procedure: Lipoaspiration — Closed Syringe Harvesting Autologous Subdermal Fat
  Arms: Lipoaspiration Arm 1
Procedure: AD-cSVF — Use of Centricyte 1000 to isolate adipose stem/stromal cells via centrifugation
  Arms: AD-cSVF Arm 2
Procedure: Normal Saline IV — Normal Saline IV containing AD-cSVF
  Arms: Normal Saline IV Arm 3

SUMMARY:
Inflammatory Bowel Disease (IBD) is a group of inflammatory conditions of the small bowel and colon. Main types include Ulcerative Colitis and Crohn's Disease. Symptoms are often difficult to distinguish except for location and nature of changes. IBD complex arises with interaction of environmental, genetic factors, immunological responses, and chronic and recurring inflammation.

Many factor appear as contributory, but no single set of issues appear to explain the process. Microbiota, intestinal wall granulation or breach, dietary, genetic predisposition all appear to factors. Treatment is often reactive or suppressive medications, neither of which appears to reverse the disease processes. This study explores the value of a complex group of adipose-derived stem/stromal cells (AD-cSVF) in the disease process.

DETAILED DESCRIPTION:
IBD often presents clinically as abdominal pain, diarrhea (with and without blood), fever, weight loss, failure to thrive, and many related symptoms. Complications of the disorders may also include anemia, skin rashes, arthritis, severe chronic fatigue, and eye inflammatory changes.

It is felt that IBD disorders may be caused by combination of environmental, immune, genetic, and bacterial factors. Results of these issues produce a chronic inflammatory disorder, in which the immune system attacks the gastrointestinal tract, perhaps directed by certain microbial antigens. The group appears not to be a pure autoimmune disease reaction, but may relate to a immunodeficiency state.

There are no medications or surgical procedures that are known to cure the diseases. Most are aimed at reduction of symptoms, maintain remissions, and try to prevent relapses. Temporary anti-inflammatory medications may improve the acute process, followed by methotrexate or thiopurine to maintain remission states. Surgery appears important in cases of perforation, abscesses, obstructions, or cancer management.

Actual occurrence is unknown, as there are more than Crohn's Disease and Ulcerative Colitis which appear related. It is estimated that more than 35,000 deaths were reported in 2010. Crohn's Disease alone appears to affect 3.2 per 1000 people in Europe and North America alone.

The usual onset of symptoms may appear before actual diagnoses are made, with typical diagnoses occurring between 15-30 years of age. Lead by abdominal pain symptoms (usually lower right quadrant) and the recurrent periods of flare and remission. Many dietary, bacterial, antimicrobials, and environmental factors receive attention, some new interest in evaluating alternative therapeutic modalities to deal of issues of immune system. Use of the immune privileged cellular agents held within the AD-cSVF is proposed to help with the inflammatory contributors as well as the modulation of inflammation which favors chronic wound healing and avascular systems. Known to provide secretory antibiotic (ll-37) contributions, some thought of pro- and anti-microbials, may prove of value in those areas specifically. Cytokine and growth factors implications at the lesion sites remain to be poorly understood, but those experienced in biocellular regenerative therapies have experienced contributions to healing and prevention of recurrences of ulcerative skin lesions.

Harvest of autologous of adipose-derived tissue stromal vascular fraction (AD-tSVF) is a proven rich resource of microvascular stem/stromal cell elements with well documented growth factor and cytokine contributors. With the advent of safe, measurable, and efficacious and reproducible numbers in a closed isolation environment, the ability to isolate and concentrate a cell-only product. This AD-cSVF is capable of reintroduction into patients, via a Normal Saline Solution, via parenteral route.

This study is intended to evaluate the safety (adverse outcomes) and efficacy of using autologous cellular therapy in cases of IBD.

ELIGIBILITY:
Inclusion Criteria:

* Patients, either sex 18 years and older with confirmed diagnosis of IBD
* Patients, either sex younger than 18 years upon approval of responsible parties and agreement of investigators
* Ability of patient to provide informed consent (or legal guardian)
* IBD diagnosed at least 6 months earlier to therapy using usual criteria
* Negative pregnancy test for women of childbearing age (menarche to menopause)

Exclusion Criteria:

* Mental incapacity that prevents adequate understanding of study and associate procedures and providing informed consent
* Severe IBD preventing tolerance of procedures needed
* Patients with impaired systemic condition, according to investigator judgment, needs immediate corticosteroid or surgical intervention
* Patients that fulfill criteria of cortico-dependency and in current treatment with corticosteroids
* Patients with history of colectomy
* Known history of alcohol, smoking dependence or additive substance abuse
* History related malignant disease - including patients participating in clinical trial with investigational drug within 6 months
* Patients with known history of allergies to any substance used in this protocol
* Pregnant or breastfeeding females
* Presence of severe concomitant disease, in investigators opinion threatens patient's well being or safety

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-11-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Safety: Inflammatory Bowel Disease | 12 months Evaluate Function and Adverse Events
  Inflammatory Bowel Disease to be addressed as occurrence or frequency of adverse event during study. Includes vital signs, complete blood count, and disease progression

SECONDARY OUTCOMES:
Efficacy: Quality of life index , Inflammatory Bowel Disease Questionnaire(IBD-QoL) | 1 month, 6 month, 1 year
  Comparison of response if it improves at least 30%
Change from Baseline in C Reactive Protein (CRP) | 0, 2 weeks, 8 weeks, 12 weeks
  Blood draw and laboratory measure of CRP as reflection of inflammatory baseline change
Efficacy: Change in Baseline of Modified Truelove-Witts Score (MTW) | 0, 4 weeks, 12 weeks
  Remission is considered if below 11, and response if it diminishes at least 30%
Efficacy: Change in Baseline in Lichtiger Index | 0, 12 weeks, 6 months
  Remission considered if reaching 0 point, and response if the score diminishes from pretreatment level

CONTACTS AND LOCATIONS:
Overall Officials: Robert W Alexander, MD, Principal Investigator — Healeon Medical Inc; Glenn C Terry, MD, Study Director — Global Alliance for Regenerative Medicine (GARM)
Locations (1):
- Regenevita LLC, Stevensville, Montana, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baumgart DC, Carding SR. Inflammatory bowel disease: cause and immunobiology. Lancet. 2007 May 12;369(9573):1627-40. doi: 10.1016/S0140-6736(07)60750-8. PMID 17499605
- [Background] Baumgart DC, Sandborn WJ. Inflammatory bowel disease: clinical aspects and established and evolving therapies. Lancet. 2007 May 12;369(9573):1641-57. doi: 10.1016/S0140-6736(07)60751-X. PMID 17499606
- [Background] Bennike T, Birkelund S, Stensballe A, Andersen V. Biomarkers in inflammatory bowel diseases: current status and proteomics identification strategies. World J Gastroenterol. 2014 Mar 28;20(12):3231-44. doi: 10.3748/wjg.v20.i12.3231. PMID 24696607
- [Background] Wang GF, Ren JA, Liu S, Chen J, Gu GS, Wang XB, Fan CG, Li JS. Clinical characteristics of non-perianal fistulating Crohn's disease in China: a single-center experience of 184 cases. Chin Med J (Engl). 2012 Jul;125(14):2405-10. PMID 22882911
- [Background] Mahadeva U, Martin JP, Patel NK, Price AB. Granulomatous ulcerative colitis: a re-appraisal of the mucosal granuloma in the distinction of Crohn's disease from ulcerative colitis. Histopathology. 2002 Jul;41(1):50-5. doi: 10.1046/j.1365-2559.2002.01416.x. PMID 12121237
- [Background] Aroniadis OC, Brandt LJ. Fecal microbiota transplantation: past, present and future. Curr Opin Gastroenterol. 2013 Jan;29(1):79-84. doi: 10.1097/MOG.0b013e32835a4b3e. PMID 23041678
- [Background] Maloy KJ, Powrie F. Intestinal homeostasis and its breakdown in inflammatory bowel disease. Nature. 2011 Jun 15;474(7351):298-306. doi: 10.1038/nature10208. PMID 21677746
- [Background] Cario E. Toll-like receptors in inflammatory bowel diseases: a decade later. Inflamm Bowel Dis. 2010 Sep;16(9):1583-97. doi: 10.1002/ibd.21282. PMID 20803699
- [Background] Coskun M. Intestinal epithelium in inflammatory bowel disease. Front Med (Lausanne). 2014 Aug 25;1:24. doi: 10.3389/fmed.2014.00024. eCollection 2014. PMID 25593900
- [Background] Feller M, Huwiler K, Schoepfer A, Shang A, Furrer H, Egger M. Long-term antibiotic treatment for Crohn's disease: systematic review and meta-analysis of placebo-controlled trials. Clin Infect Dis. 2010 Feb 15;50(4):473-80. doi: 10.1086/649923. PMID 20067425
- [Background] Mowat C, Cole A, Windsor A, Ahmad T, Arnott I, Driscoll R, Mitton S, Orchard T, Rutter M, Younge L, Lees C, Ho GT, Satsangi J, Bloom S; IBD Section of the British Society of Gastroenterology. Guidelines for the management of inflammatory bowel disease in adults. Gut. 2011 May;60(5):571-607. doi: 10.1136/gut.2010.224154. PMID 21464096
- [Background] Charlebois A, Rosenfeld G, Bressler B. The Impact of Dietary Interventions on the Symptoms of Inflammatory Bowel Disease: A Systematic Review. Crit Rev Food Sci Nutr. 2016 Jun 10;56(8):1370-8. doi: 10.1080/10408398.2012.760515. PMID 25569442
- [Background] Colman RJ, Rubin DT. Fecal microbiota transplantation as therapy for inflammatory bowel disease: a systematic review and meta-analysis. J Crohns Colitis. 2014 Dec;8(12):1569-81. doi: 10.1016/j.crohns.2014.08.006. Epub 2014 Sep 13. PMID 25223604
- [Background] Gilardi D, Fiorino G, Genua M, Allocca M, Danese S. Complementary and alternative medicine in inflammatory bowel diseases: what is the future in the field of herbal medicine? Expert Rev Gastroenterol Hepatol. 2014 Sep;8(7):835-46. doi: 10.1586/17474124.2014.917954. Epub 2014 May 12. PMID 24813226
- [Background] Langhorst J, Wulfert H, Lauche R, Klose P, Cramer H, Dobos GJ, Korzenik J. Systematic review of complementary and alternative medicine treatments in inflammatory bowel diseases. J Crohns Colitis. 2015 Jan;9(1):86-106. doi: 10.1093/ecco-jcc/jju007. Epub 2014 Nov 28. PMID 25518050
- [Background] Dave M, Mehta K, Luther J, Baruah A, Dietz AB, Faubion WA Jr. Mesenchymal Stem Cell Therapy for Inflammatory Bowel Disease: A Systematic Review and Meta-analysis. Inflamm Bowel Dis. 2015 Nov;21(11):2696-707. doi: 10.1097/MIB.0000000000000543. PMID 26230863
- [Background] Ghouri YA, Richards DM, Rahimi EF, Krill JT, Jelinek KA, DuPont AW. Systematic review of randomized controlled trials of probiotics, prebiotics, and synbiotics in inflammatory bowel disease. Clin Exp Gastroenterol. 2014 Dec 9;7:473-87. doi: 10.2147/CEG.S27530. eCollection 2014. PMID 25525379
- [Background] Thomas S, Baumgart DC. Targeting leukocyte migration and adhesion in Crohn's disease and ulcerative colitis. Inflammopharmacology. 2012 Feb;20(1):1-18. doi: 10.1007/s10787-011-0104-6. Epub 2011 Dec 20. PMID 22205271
- [Background] Del Pinto R, Pietropaoli D, Chandar AK, Ferri C, Cominelli F. Association Between Inflammatory Bowel Disease and Vitamin D Deficiency: A Systematic Review and Meta-analysis. Inflamm Bowel Dis. 2015 Nov;21(11):2708-17. doi: 10.1097/MIB.0000000000000546. PMID 26348447
- [Background] Dessein R, Chamaillard M, Danese S. Innate immunity in Crohn's disease: the reverse side of the medal. J Clin Gastroenterol. 2008 Sep;42 Suppl 3 Pt 1:S144-7. doi: 10.1097/MCG.0b013e3181662c90. PMID 18806708
- [Background] Marks DJ, Rahman FZ, Sewell GW, Segal AW. Crohn's disease: an immune deficiency state. Clin Rev Allergy Immunol. 2010 Feb;38(1):20-31. doi: 10.1007/s12016-009-8133-2. PMID 19437144
- [Background] Casanova JL, Abel L. Revisiting Crohn's disease as a primary immunodeficiency of macrophages. J Exp Med. 2009 Aug 31;206(9):1839-43. doi: 10.1084/jem.20091683. Epub 2009 Aug 17. PMID 19687225
- [Background] Lalande JD, Behr MA. Mycobacteria in Crohn's disease: how innate immune deficiency may result in chronic inflammation. Expert Rev Clin Immunol. 2010 Jul;6(4):633-41. doi: 10.1586/eci.10.29. PMID 20594136
- [Background] Yamamoto-Furusho JK, Korzenik JR. Crohn's disease: innate immunodeficiency? World J Gastroenterol. 2006 Nov 14;12(42):6751-5. doi: 10.3748/wjg.v12.i42.6751. PMID 17106921
- [Background] Molodecky NA, Soon IS, Rabi DM, Ghali WA, Ferris M, Chernoff G, Benchimol EI, Panaccione R, Ghosh S, Barkema HW, Kaplan GG. Increasing incidence and prevalence of the inflammatory bowel diseases with time, based on systematic review. Gastroenterology. 2012 Jan;142(1):46-54.e42; quiz e30. doi: 10.1053/j.gastro.2011.10.001. Epub 2011 Oct 14. PMID 22001864
- [Background] Trikudanathan G, Venkatesh PG, Navaneethan U. Diagnosis and therapeutic management of extra-intestinal manifestations of inflammatory bowel disease. Drugs. 2012 Dec 24;72(18):2333-49. doi: 10.2165/11638120-000000000-00000. PMID 23181971
- [Background] Braat H, Peppelenbosch MP, Hommes DW. Immunology of Crohn's disease. Ann N Y Acad Sci. 2006 Aug;1072:135-54. doi: 10.1196/annals.1326.039. PMID 17057196
- [Background] Henckaerts L, Figueroa C, Vermeire S, Sans M. The role of genetics in inflammatory bowel disease. Curr Drug Targets. 2008 May;9(5):361-8. doi: 10.2174/138945008784221161. PMID 18473763
- [Background] Marks DJ, Harbord MW, MacAllister R, Rahman FZ, Young J, Al-Lazikani B, Lees W, Novelli M, Bloom S, Segal AW. Defective acute inflammation in Crohn's disease: a clinical investigation. Lancet. 2006 Feb 25;367(9511):668-78. doi: 10.1016/S0140-6736(06)68265-2. PMID 16503465
- [Background] Clevers H. Inflammatory bowel disease, stress, and the endoplasmic reticulum. N Engl J Med. 2009 Feb 12;360(7):726-7. doi: 10.1056/NEJMcibr0809591. No abstract available. PMID 19213688
- [Background] Elson CO, Cong Y, Weaver CT, Schoeb TR, McClanahan TK, Fick RB, Kastelein RA. Monoclonal anti-interleukin 23 reverses active colitis in a T cell-mediated model in mice. Gastroenterology. 2007 Jun;132(7):2359-70. doi: 10.1053/j.gastro.2007.03.104. Epub 2007 Apr 13. PMID 17570211
- [Background] Naser SA, Sagramsingh SR, Naser AS, Thanigachalam S. Mycobacterium avium subspecies paratuberculosis causes Crohn's disease in some inflammatory bowel disease patients. World J Gastroenterol. 2014 Jun 21;20(23):7403-15. doi: 10.3748/wjg.v20.i23.7403. PMID 24966610
- [Background] Cenac N, Andrews CN, Holzhausen M, Chapman K, Cottrell G, Andrade-Gordon P, Steinhoff M, Barbara G, Beck P, Bunnett NW, Sharkey KA, Ferraz JG, Shaffer E, Vergnolle N. Role for protease activity in visceral pain in irritable bowel syndrome. J Clin Invest. 2007 Mar;117(3):636-47. doi: 10.1172/JCI29255. Epub 2007 Feb 15. PMID 17304351
- [Background] Hara AK, Leighton JA, Heigh RI, Sharma VK, Silva AC, De Petris G, Hentz JG, Fleischer DE. Crohn disease of the small bowel: preliminary comparison among CT enterography, capsule endoscopy, small-bowel follow-through, and ileoscopy. Radiology. 2006 Jan;238(1):128-34. doi: 10.1148/radiol.2381050296. PMID 16373764
- [Background] Broome U, Bergquist A. Primary sclerosing cholangitis, inflammatory bowel disease, and colon cancer. Semin Liver Dis. 2006 Feb;26(1):31-41. doi: 10.1055/s-2006-933561. PMID 16496231
- [Background] Kristo I, Stift A, Bergmann M, Riss S. Surgical recurrence in Crohn's disease: Are we getting better? World J Gastroenterol. 2015 May 28;21(20):6097-100. doi: 10.3748/wjg.v21.i20.6097. PMID 26034346
- [Background] Joos S, Brinkhaus B, Maluche C, Maupai N, Kohnen R, Kraehmer N, Hahn EG, Schuppan D. Acupuncture and moxibustion in the treatment of active Crohn's disease: a randomized controlled study. Digestion. 2004;69(3):131-9. doi: 10.1159/000078151. Epub 2004 Apr 26. PMID 15114043
- [Background] Smart HL, Mayberry JF, Atkinson M. Alternative medicine consultations and remedies in patients with the irritable bowel syndrome. Gut. 1986 Jul;27(7):826-8. doi: 10.1136/gut.27.7.826. PMID 3755416
- [Background] Axelrad JE, Lichtiger S, Yajnik V. Inflammatory bowel disease and cancer: The role of inflammation, immunosuppression, and cancer treatment. World J Gastroenterol. 2016 May 28;22(20):4794-801. doi: 10.3748/wjg.v22.i20.4794. PMID 27239106
- [Result] Walker MM, Murray JA. An update in the diagnosis of coeliac disease. Histopathology. 2011 Aug;59(2):166-79. doi: 10.1111/j.1365-2559.2010.03680.x. Epub 2010 Nov 3. PMID 21054494